CLINICAL TRIAL: NCT05095727
Title: A Phase 1/2, Adaptive, Open-label, Single Ascending Dose to Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of mRNA-3745 in Participants With Glycogen Storage Disease Type 1a (GSD1a), Followed by an Open-label Extension
Brief Title: A Study of mRNA-3745 in Adult and Pediatric Participants With Glycogen Storage Disease Type 1a (GSD1a)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-3745-P102; 2022-502963-39-00 (Registry Identifier: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2021-10-04; First posted 2021-10-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Glycogen Storage Disease
Keywords: Glycogen storage disease type 1a; GSD1a; Von Gierke disease; Glucose metabolism disorder; Genetic disorder; Autosomal recessive disorder; messenger RNA; mRNA; Pediatric
MeSH Terms: conditions — Glycogen Storage Disease; Glycogen Storage Disease Type I; Glucose Metabolism Disorders; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAD: mRNA-3745 (Experimental): Participants will receive a single intravenous (IV) dose of mRNA-3745 on Day 1 in an inpatient setting. Participants that are/have been enrolled in the study and receive an administration of mRNA-3745 may also enroll in one of the MAD cohorts. The first MAD dose must occur at least 21 days after the SAD dose.
  Interventions: Drug: mRNA-3745
- MAD: mRNA-3745 (Experimental): Participants will receive multiple IV doses of mRNA-3745 in an inpatient setting. Participants will have the option to continue treatment in the OLE.
  Interventions: Drug: mRNA-3745

INTERVENTIONS:
Drug: mRNA-3745 — Sterile frozen liquid dispersion for injection

SUMMARY:
The main goal of this trial is to evaluate the safety and tolerability of mRNA-3745 via intravenous (IV) administration in adult and pediatric participants with GSD1a.

DETAILED DESCRIPTION:
The study includes a single ascending dose (SAD) stage and a multiple ascending dose (MAD) stage. Participants enrolled in the MAD stage have the option to continue treatment in an open-label extension (OLE) period that will assess long-term safety and clinical activity of mRNA-3745.

ELIGIBILITY:
Inclusion Criteria:

* Documented GSD1a with confirmation of biallelic gene encoding glucose-6-phosphatase-α (G6PC) mutations by genetic testing.
* Absence of hospitalization for hypoglycemia in the 4 weeks prior to Screening

Exclusion Criteria:

* Solid organ transplant
* Received gene therapy for GSD1a
* Presence of liver adenoma >5 centimeters (cm) in size
* Diagnosis of type 1 or type 2 diabetes mellitus
* Presence of liver adenoma with growth of >2 cm or >5 newly diagnosed liver adenomas, in the previous 2 years

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and TEAEs Leading to Treatment Discontinuation | Day 1 up to approximately 3.5 years

SECONDARY OUTCOMES:
Number of Participants Not Experiencing Hypoglycemia During Fasting Challenges | Baseline through up to Week 32
  Hypoglycemia is defined as blood glucose <60 milligrams (mg)/deciliter (dL) (3.3 millimoles [mmol]/liter [L]) and/or symptoms of hypoglycemia.
Change From Baseline of Area Under the Effect Curve (AUEC) of Blood Glucose and Lactate During Fasting Challenges | Baseline through up to Week 32
Change From Baseline in Time to Hypoglycemia During Fasting Challenges | Baseline through up to Week 32
Change From Baseline in Maximum Effect (Emax) During Fasting Challenges | Baseline through up to Week 32
SAD only: Maximum Observed Concentration (Cmax) of Messenger Ribonucleic Acid (mRNA) and Lipid Nanoparticle (LNP) | Pre-infusion, during infusion, at the end of infusion (EOI) and post-infusion on Day 1 up to Week 52
SAD only: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUC0-t) of mRNA and LNP | Pre-infusion, during infusion, at EOI and post-infusion on Day 1 up to Week 52
Change From Baseline in Metabolic Biomarkers of GSD1a | Baseline through up to approximately 6.5 years
MAD only: Maximum Observed Concentration at Steady State (Cmax,ss) of mRNA and LNP | Pre-infusion, during infusion, at the EOI and post-infusion on Day 1 up to Week 52

CONTACTS AND LOCATIONS:
Locations (16):
- United States (8):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - Stollery Children's Hospital University of Alberta, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
- France (2):
  - AP-HP - Hôpital Antoine Béclère, Clamart
  - CHRU Tours - Hopital Clocheville, Tours
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw, Poland
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga

REFERENCES:
- [Background] Cao J, Choi M, Guadagnin E, Soty M, Silva M, Verzieux V, Weisser E, Markel A, Zhuo J, Liang S, Yin L, Frassetto A, Graham AR, Burke K, Ketova T, Mihai C, Zalinger Z, Levy B, Besin G, Wolfrom M, Tran B, Tunkey C, Owen E, Sarkis J, Dousis A, Presnyak V, Pepin C, Zheng W, Ci L, Hard M, Miracco E, Rice L, Nguyen V, Zimmer M, Rajarajacholan U, Finn PF, Mithieux G, Rajas F, Martini PGV, Giangrande PH. mRNA therapy restores euglycemia and prevents liver tumors in murine model of glycogen storage disease. Nat Commun. 2021 May 25;12(1):3090. doi: 10.1038/s41467-021-23318-2. PMID 34035281